CLINICAL TRIAL: NCT04339998
Title: Assessment of Exam Findings in Coronavirus Disease 2019 (COVID-19) With Point-of-Care Ultrasonography (POCUS)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: GIM-2020-28740
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Infection; COVID; Covid-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Suspected or Confirmed COVID-19: Patients 18 years of age and older under investigation for COVID-19 and those patients that are positive for COVID-19 at University of Minnesota Medical Center and Bethesda Hospital. Informed consent will be obtained from the patient or decision maker prior to study inclusion
  Interventions: Diagnostic Test: Point-of-Care Ultrasonography (POCUS)

INTERVENTIONS:
Diagnostic Test: Point-of-Care Ultrasonography (POCUS) — The POCUS exam of the heart will capture 2 standard views commonly used to assess general cardiac function at the point of care. The details of POCUS views and exam findings of interest are outline below:
  Pulmonary POCUS Evaluation:
  1. B lines: absent (< 3 lines), present (> 3 lines), fused
  2. Consolidation: yes or no
     a. Bilateral: yes or no
  3. Pleural Effusion: yes or no
  4. Other pleural abnormalities: yes or no Score each finding based on degree of abnormalities and number of sites with abnormalities
  Cardiac POCUS Evaluation:
  1. Parasternal long axis
  2. Parasternal short axis
     1. Qualitative LVEF: Normal, hyperdynamic, mild-moderately depressed, severely depressed
     2. EPSS (E-point septal separation): normal (<10 mm), abnormal (>10 mm)
     3. Left ventricular (LV) mass approximation by septal thickness
     4. Left Ventricular Chamber Size by internal diameter at diastole

SUMMARY:
Specific Aims:

1. The investigators will prospectively evaluate and analyze changes in the appearance of the lungs and heart through serial acquisition of focused point-of-care ultrasound images in a cohort of patients with or under investigation for COVID-19.
2. The investigators will correlate changes noted in ultrasound with clinical course and diagnostic evaluation to ascertain whether changes on ultrasound could improve care through earlier diagnosis or identification of patients at high risk of disease progression.

DETAILED DESCRIPTION:
The investigators will perform a descriptive study aimed at identifying the cardiopulmonary ultrasound features in patients with or under investigation for COVID-19.

The study will take place at two sites: University of Minnesota Medical Center (UMMC) and Bethesda Hospital. At UMMC, a tertiary care center, clinicians will recruit and evaluate patients with or under investigation for COVID-19. At Bethesda clinicians will recruit and evaluate patients with a confirmed diagnosis of COVID-19 as demonstrated by a positive PT-PCR.

POCUS exams will be performed in a cohort of 200-500 patients with or under investigation for COVID-19. Serial ultrasound examinations will be performed every 48-72 hours until discharge, death, or study completion. Participants will undergo POCUS at enrollment by their treating physicians. Inquiry into study enrollment will be performed over the phone rather than in person, given the current scarcity of PPE and the added use that would occur with in-person enrollment.

ELIGIBILITY:
Inclusion Criteria:

* patients under investigation for COVID-19
* patients that are positive for COVID-19 at UMMC and Bethesda

Exclusion Criteria:

- ultrasound contraindication such as overlying skin wound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older under investigation for COVID-19 and those patients that are positive for COVID-19 at UMMC and Bethesda. Informed consent will be obtained from the patient or decision maker prior to study inclusion.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
POCUS Score - Lungs | up to 14 days
  POCUS is a 6-point scale evaluating the degree of abnormalities and number of sites with abnormalities in ultrasound images of the lungs. Higher scores indicate greater malady.
  Pulmonary POCUS Evaluation:
  1. B lines: absent (< 3 lines), present (> 3 lines), fused
  2. Consolidation: yes or no
     a. Bilateral: yes or no
  3. Pleural Effusion: yes or no
  4. Other pleural abnormalities: yes or no
  Score each finding based on degree of abnormalities and number of sites with abnormalities
POCUS Score - Heart | up to 14 days
  POCUS is a 6-point scale evaluating the degree of abnormalities and number of sites with abnormalities in ultrasound images of the heart. Higher scores indicate greater malady.
  Cardiac POCUS Evaluation:
  1. Parasternal long axis
  2. Parasternal short axis
     1. Qualitative LVEF: Normal, hyperdynamic, mild-moderately depressed, severely depressed
     2. EPSS (E-point septal separation): normal (<10 mm), abnormal (>10 mm)
     3. Left ventricular (LV) mass approximation by septal thickness
     4. Left Ventricular Chamber Size by internal diameter at diastole
  Score each finding based on degree of abnormalities and number of sites with abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Yocum, MD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Medical Center (UMMC), Minneapolis, Minnesota
  - M Health Fairview Bethesda Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided